CLINICAL TRIAL: NCT05979025
Title: Factors Predicting the Need for Endoscopic Intervention in Non-variceal Upper Gastrointestinal Bleeding
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Numan Aydın, Medical Doctor, Ankara City Hospital Bilkent
Other Study IDs: AnkaraCHBilkent-NA-TEZ
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Acute Upper Gastrointestinal Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastrointestinal system bleedings are medical emergencies and the most common cause of hospital admissions related to digestive system diseases. Gastrointestinal system bleedings are a frequently encountered condition and one of the significant reasons leading to morbidity, mortality, and medical care costs. For acute upper gastrointestinal system bleedings, the annual hospital admission incidence in the United States is approximately 67 per 100,000 adults, making it more common than lower gastrointestinal system bleedings. Approximately 80% of acute upper gastrointestinal system bleedings are attributed to non-variceal causes. Endoscopy is an invasive procedure used for diagnosis and treatment in upper gastrointestinal system bleedings. . In recent years, there has been an increase in endoscopy and endoscopic treatment rates. Except for variceal bleedings, most upper gastrointestinal system bleedings stop without the need for endoscopic intervention. However, some patients require endoscopic intervention and identifying this high-risk group, prone to recurrent bleeding, through non-invasive tests is crucial. In investigators' prospective study, researcher aimed to facilitate the identification of patients who require intervention and undergo endoscopic intervention (e.g., epinephrine injection, hemoclips, thermal coagulation, argon plasma coagulation, etc.) among those who underwent endoscopy within the first 24 hours after admission to the hospital's emergency department with a diagnosis of non-variceal acute upper gastrointestinal system bleeding. Investigators sought to achieve this by determining the relevant parameters related to their clinical and laboratory findings, comorbidities, and demographic characteristics at the time of admission. This approach aims to reduce hospital admissions, hospital stay, and costs, and particularly to minimize interventional procedures during seizures and decrease complications.As of August 2022, patients who applied to the Ankara Bilkent City Hospital emergency department were followed up.

DETAILED DESCRIPTION:
Gastrointestinal system bleedings are medical emergencies and the most common cause of hospital admissions related to digestive system diseases. Gastrointestinal system bleedings are a frequently encountered condition and one of the significant reasons leading to morbidity, mortality, and medical care costs. For acute upper gastrointestinal system bleedings, the annual hospital admission incidence in the United States is approximately 67 per 100,000 adults, making it more common than lower gastrointestinal system bleedings. A decrease in the incidence of non-variceal acute upper gastrointestinal system bleeding has been observed compared to previous years, which is believed to be associated with an increase in the use of proton pump inhibitors (PPIs), eradication of Helicobacter pylori (H. pylori), and advancements in endoscopic treatment. Approximately 80% of acute upper gastrointestinal system bleedings are attributed to non-variceal causes.

Endoscopy is an invasive procedure used for diagnosis and treatment in upper gastrointestinal system bleedings. In recent years, there has been an increase in endoscopy and endoscopic treatment rates. Previous studies have identified higher mortality rates, around 5-10% for bleeding due to peptic ulcers, and approximately 15% for esophageal variceal bleedings. The development of modern endoscopy has led to significant advancements in various therapeutic techniques. Mortality related to all causes of upper gastrointestinal system bleedings has declined due to advancements in treatment. In recent years, there has been a decrease in hospitalization duration and mortality, but the total economic burden has significantly increased.

Except for variceal bleedings, most upper gastrointestinal system bleedings stop without the need for endoscopic intervention. However, some patients require endoscopic intervention and identifying this high-risk group, prone to recurrent bleeding, through non-invasive tests is crucial. In cases where endoscopic treatment is insufficient, surgical or interventional radiology procedures such as embolization may be necessary. Endoscopic treatment has led to a reduction in the need for surgery and blood transfusions in patients presenting with upper gastrointestinal system bleeding. The goal of treatment is to prevent complications and deaths. Determining the need for treatment for a patient is clinically and practically easier than predicting who will die or re-bleed.

Gastrointestinal bleedings can lead to various clinical scenarios due to multiple lesion types, and they can occur from any part of the gastrointestinal system, either overtly or covertly. Upper gastrointestinal bleedings are approximately 5 times more common than lower gastrointestinal bleedings. Several scoring systems, such as Glasgow-Blatchford, Rockall, AIMS65, have been developed to predict the need for endoscopic intervention, risk of re-bleeding, and 30-day mortality in non-variceal bleedings.

Emergency upper gastrointestinal endoscopy is performed within the first 12 hours in high-risk patients who present to the hospital's emergency department with acute upper gastrointestinal system bleeding. However, it may not always be feasible to adhere to this timeframe, and endoscopy can be performed up to 24 hours after appropriate resuscitation, depending on the expertise of the personnel.

In investigators' prospective study, researcher aimed to facilitate the identification of patients who require intervention and undergo endoscopic intervention (e.g., epinephrine injection, hemoclips, thermal coagulation, argon plasma coagulation, etc.) among those who underwent endoscopy within the first 24 hours after admission to the hospital's emergency department with a diagnosis of non-variceal acute upper gastrointestinal system bleeding. Investigators sought to achieve this by determining the relevant parameters related to their clinical and laboratory findings, comorbidities, and demographic characteristics at the time of admission. This approach aims to reduce hospital admissions, hospital stay, and costs, and particularly to minimize interventional procedures during seizures and decrease complications. As of August 2022, patients who applied to the Ankara Bilkent City Hospital emergency department were followed up.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to our hospital with a diagnosis of non-variceal upper gastrointestinal bleeding
* Patients who undergo endoscopy within the first 24 hours after hospital admission

Exclusion Criteria:

* Patients who have variceal bleeding
* Lower gastrointestinal system bleeding
* Individuals who are under the age of 18
* Patients who do not undergo endoscopy within the first 24 hours after hospital admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are 18 years of age and older and present to our hospital with a diagnosis of non-variceal upper gastrointestinal bleeding, among whom endoscopy is performed within the first 24 hours after hospital admission
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-07-29 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Endoscopic intervention | First 24 hours after hospital admission
  Mechanical treatment (eg hemoclips, tape, etc.), injection therapy (eg epinephrine etc.), thermal coagulation (eg heater probe etc.)

SECONDARY OUTCOMES:
İntensive care hospitalization | 30 days after admission to hospital
  Intensive care unit (ICU) admission of patients presenting to the hospital due to non-variceal upper gastrointestinal system bleeding either at the time of admission or within 30 days after hospitalization for any reason.
Mortality | 30 days after admission to hospital
  Death within 30 days of hospital admission with non-variceal upper gastrointestinal bleeding
Rebleeding | 30 days after admission to hospital
  Rebleeding within 30 days of hospital admission with non-variceal upper gastrointestinal bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wuerth BA, Rockey DC. Changing Epidemiology of Upper Gastrointestinal Hemorrhage in the Last Decade: A Nationwide Analysis. Dig Dis Sci. 2018 May;63(5):1286-1293. doi: 10.1007/s10620-017-4882-6. Epub 2017 Dec 27. PMID 29282637
- [Result] Abougergi MS, Travis AC, Saltzman JR. The in-hospital mortality rate for upper GI hemorrhage has decreased over 2 decades in the United States: a nationwide analysis. Gastrointest Endosc. 2015 Apr;81(4):882-8.e1. doi: 10.1016/j.gie.2014.09.027. Epub 2014 Dec 5. PMID 25484324
- [Result] Masaoka T, Suzuki H, Hori S, Aikawa N, Hibi T. Blatchford scoring system is a useful scoring system for detecting patients with upper gastrointestinal bleeding who do not need endoscopic intervention. J Gastroenterol Hepatol. 2007 Sep;22(9):1404-8. doi: 10.1111/j.1440-1746.2006.04762.x. PMID 17716345
- [Result] Chen IC, Hung MS, Chiu TF, Chen JC, Hsiao CT. Risk scoring systems to predict need for clinical intervention for patients with nonvariceal upper gastrointestinal tract bleeding. Am J Emerg Med. 2007 Sep;25(7):774-9. doi: 10.1016/j.ajem.2006.12.024. PMID 17870480
- [Result] Lanas A, Dumonceau JM, Hunt RH, Fujishiro M, Scheiman JM, Gralnek IM, Campbell HE, Rostom A, Villanueva C, Sung JJY. Non-variceal upper gastrointestinal bleeding. Nat Rev Dis Primers. 2018 Apr 19;4:18020. doi: 10.1038/nrdp.2018.20. PMID 29671413
- [Result] Kamboj AK, Hoversten P, Leggett CL. Upper Gastrointestinal Bleeding: Etiologies and Management. Mayo Clin Proc. 2019 Apr;94(4):697-703. doi: 10.1016/j.mayocp.2019.01.022. PMID 30947833
- [Result] Wilkins T, Wheeler B, Carpenter M. Upper Gastrointestinal Bleeding in Adults: Evaluation and Management. Am Fam Physician. 2020 Mar 1;101(5):294-300. PMID 32109037
- [Result] Rockey DC. Gastrointestinal bleeding. Gastroenterol Clin North Am. 2005 Dec;34(4):581-8. doi: 10.1016/j.gtc.2005.08.002. PMID 16303571
- [Result] Lakatos L, Gonczi L, Lontai L, Izbeki F, Patai A, Racz I, Gasztonyi B, Varga-Szabo L, Ilias A, Lakatos PL. Incidence, Predictive Factors, Clinical Characteristics and Outcome of Non-variceal Upper Gastrointestinal Bleeding - A Prospective Population-based Study from Hungary. J Gastrointestin Liver Dis. 2021 Sep 21;30(3):327-333. doi: 10.15403/jgld-3495. PMID 34375379